CLINICAL TRIAL: NCT06034613
Title: The Effects and Mechanisms of Mindfulness Intervention for Emotional Distress: Daily Interventions and Daily Assessments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xinghua Liu, Director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20230830
Record Dates: First submitted 2023-09-01; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Emotional Distress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mindfulness intervention group (Experimental): provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression and other emotions, the source of anxiety, depression and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Interventions: Behavioral: internet-based mindfulness intervention for emotional distress(iMIED）

INTERVENTIONS:
Behavioral: internet-based mindfulness intervention for emotional distress(iMIED） — The iMIED program integrates the rationales and practices from the UP and MBIs. Formal mindfulness exercises (e.g., body scan, mindful breathing, and mindful stretching) and informal mindfulness practices (e.g., mindful tooth brushing) were adapted from MBIs. In addition, the iMIED program selected several important tasks from the UP, like practicing tolerating uncomfortable feelings by interoceptive exposure practices (e.g., rapid breathing), identifying avoidant behaviors and emotion-driven behaviors and reducing them step by step, identifying common maladaptive automatic thoughts (e.g., overestimating probability and catastrophizing), and using the above strategies in daily life by completing challenging tasks. In total, it took about 30 min per day to finish all the tasks. The program lasted for 49 days.

SUMMARY:
This clinical trial seeks to uncover the mechanisms behind the effectiveness of mindfulness-based interventions in reducing emotional distress. Using daily diaries to measure both mediating and outcome variables, the study examines whether these mechanisms precede changes in outcomes. It focuses on the Mindfulness Intervention for Emotional Distress program, which includes four strategies. The current study plans to employ a within-subjects design with daily questionnaires over 63 days, before, during and after the intervention. The aim is to gain insights into how mindfulness interventions work in alleviating emotional distress.

DETAILED DESCRIPTION:
An abundance of research studies has demonstrated the potential efficacy of mindfulness-based interventions in alleviating emotional distress among individuals. However, the underlying mechanisms driving these effects have remained largely unknown. Furthermore, many of the mechanistic investigations have not taken into account the temporal precedence, where changes in mechanisms occur prior to changes in outcome variables.

To address these gaps, this clinical trial aims to enhance our understanding of the mechanisms behind mindfulness-based interventions for emotional distress. By employing a daily diary approach to measure both mediating and outcome variables, investigators seek to rigorously examine whether the proposed mediating variables adhere to the criterion of temporal precedence. Additionally, utilizing daily diaries allows for the collection of extensive individual-level data. This approach also permits a network analysis perspective to explore the roles of various mechanistic variables in the context of mitigating emotional distress.

The present study focuses on the Mindfulness Intervention for Emotional Distress program (liu, in press), comprising four key strategies: 1) Engaging in life to restore a sense of normalcy; 2) Enhancing distress tolerance; 3) Reducing excessive emotional reactivity; 4) Cultivating cognitive flexibility by treating thoughts as mere mental events. Through the implementation of daily diaries, investigators aim to uncover the mechanistic workings of these four strategies.

The current study plans to employ a within-subjects design, with participants all receiving mindfulness intervention. They are required to complete daily measurement questionnaires during the week prior to intervention, throughout the intervention period, and for a week following the intervention. The measurement period spans a total of 63 days.

Through this study design, investigators aim to gain valuable insights into the mechanisms underpinning the effectiveness of mindfulness interventions in alleviating emotional distress.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with scores greater than 21 on the Kessler Psychological Distress Scale.

Exclusion Criteria:

* Subjects who could not access the Internet.
* Subjects with insufficient Chinese ability.
* Subjects who have participated in mindfulness-based projects for more than 6 weeks before, and / or the current frequency of meditation practice is more than once a week.
* Patients with schizophrenia or psychotic affective disorder, current organic mental disorder, substance abuse disorder and generalized developmental disorder.
* Subjects at risk of suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-18 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Daily changes of mindfulness | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  The Daily Mindfulness Response Scale measures the frequency with which one returns to a nonjudgmental and unconditionally receptive present moment awareness during the day. Each item is rated on a scale ranging from 1 (rarely)to10(often).
  scores range from 4 to 40, with higher scores indicating higher levels of mindful responding
Daily changes of engaging in everyday life | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Self-developed questionnaire, measuring to what extent individuals put efforts and time in engaging in everyday life (e.g., work, social, leisure...), 6 items, scores range from 6 to 54, with higher scores indicating higher levels of engaging in everyday life
Daily changes of distress tolerance | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  measured by Daily distress tolerance scale, four items, scores range from 4 to 20, with higher scores indicating higher levels of distress tolerance.
Daily changes of excessive emotion behaviors | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  self-developed scale, measuring to what extent individuals use excessive emotion behaviors to control aversive feelings and emotions, 4 items, scores range from 4 to 20, with higher scores indicating higher levels of using excessive emotion behaviors.
Daily changes of cognitive flexibility/treating thoughts as thoughts | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  self-developed questionnaire, measuring to what extent individuals could treat thoughts as psychological phenomenon rather than facts, 4 items, scores range from 4 to 20, with higher scores indicating higher levels of cognitive flexibility.
daily changes of anxiety | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Daily Anxiety Severity and Impairment Scale,5 items, scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
daily changes of depression | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Daily Depression Severity and Impairment Scale,5 items, scores range from 0 to 20, with higher scores indicating higher levels of depression.
Daily changes of positive and negative affect | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Daily positive and negative affect were measured using the 10-itemInternational Positive and Negative Affect Schedule-Short Form Scale. Scores range from 5 to 25, with higher scores indicating higher levels of positive/negative affect.
daily stress | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Daily perceived stress was assessed with the previously validated four-item version of the Perceived Stress Scale, The PSS measures the degree to which situations in one's life are evaluated as stressful (e.g., "Today, to what extent did you feel confident about your ability to handle your personal problems?"). Participants rated the accuracy of the items using a scale ranging from 1 (very little)to 10 (very much). scores range from 4 to 40.

SECONDARY OUTCOMES:
daily stressors | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Daily stressor exposure was measured with 1 item, 0 = no, 1 = yes
pre-post changes of Five Facet Mindfulness Questionnaire | 1 week before the intervention, 1week after the intervention
  The Five Facet Mindfulness Questionnaire is a self-reported questionnaire measuring mindfulness levels. Scores range from 39 to 195, with higher scores indicating higher levels of mindfulness.
pre-post changes of Chinese Perceived Stress Scale | 1 week before the intervention, 1week after the intervention
  The Chinese Perceived Stress Scale is a self-reported questionnaire measuring stress. Scores range from 0 to 56, with higher scores indicating higher levels of stress
pre-post changes of 10-item Kessler Psychological Distress Scale | 1 week before the intervention, 1week after the intervention
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress.
pre-post changes of the Overall Anxiety Severity and Impairment Scale | 1 week before the intervention, 1week after the intervention
  The Overall Anxiety Severity and Impairment Scale is a self-reported questionnaire measuring anxiety. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
pre-post changes of the Overall Depression Severity and Impairment Scale | 1 week before the intervention, 1week after the intervention
  The Overall Depression Severity and Impairment Scale is a self-reported questionnaire measuring depression. Scores range from 0 to 20, with higher scores indicating higher levels of depression.
pre-post changes of Patient Health Questionnaire during the intervention | 1 week before the intervention, 1week after the intervention
  The Patient Health Questionnaire is a self-reported questionnaire measuring the degree of being troubled by various common physical symptoms. Scores range from 0 to 30.0~4 scores: no physical symptoms; 5~9 scores: mild physical symptoms; 10~14 scores: moderate physical symptoms; 15~30 scores: severe physical symptoms.
pre-post changes of Distress Tolerance Scale | 1 week before the intervention, 1week after the intervention
  Distress Tolerance Scale is used to measure Distress Tolerance. Scores range from 5 to 75, with higher scores indicating higher levels of Distress Tolerance.
pre-post changes of Beck Anxiety Inventory | 1 week before the intervention, 1week after the intervention
  Beck Anxiety Inventory is a self-reported questionnaire measuring Anxiety level.Scores range from 0 to 63, with higher scores indicating higher levels of Anxiety.
pre-post changes of Beck Depression Inventory | 1 week before the intervention, 1week after the intervention
  Beck Depression Inventory is a self-reported questionnaire measuring depression level.Scores range from 0 to 63, with higher scores indicating higher levels of depression.
pre-post changes of Athens Insomnia Scale | 1 week before the intervention, 1week after the intervention
  The Athens Insomnia Scale is a self-reported questionnaire measuring sleepy quality. Scores range from 0 to 24, with lower scores indicating higher levels of sleep quality.
pre-post changes of engaging in everyday life | 1 week before the intervention, 1week after the intervention
  The Chinese version of the Likert 5-point self-administered scale contains five dimensions, including sleep, diet, socialization, work and study, and other aspects, with a total of 15 entries, and the higher the total score indicates the worse the state of life compared with the surrounding people. The internal consistency reliability of the scale was 0.895, and the results of factor analysis and convergent validity analysis were good.
pre-post changes of treating thoughts as thoughts/cognitive flexibility | 1 week before the intervention, 1week after the intervention
  The questionnaire has 1 dimension and contains 6 items on a five-point Likert scale (1=completely compliant, 5=completely non-compliant), with higher scores indicating higher ability to treat ideas as ideas.
pre-post changes of the Brief Experiential Avoidance Questionnaire | 1 week before the intervention, 1week after the intervention
  Chinese version of the Brief Experiential Avoidance Questionnaire scale is used to measure Experiential Avoidance.Scores range from 15 to 90, with higher scores indicating higher levels of experiential avoidance.
pre-post changes of the Rumination sub-scale | 1 week before the intervention, 1week after the intervention
  12 items from the Rumination-Reflection Questionnaire, the Rumination subscale. Total scores range from 5 to 60, with higher scores indicating higher levels of rumination.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University

IPD SHARING:
Plan to Share IPD: No